CLINICAL TRIAL: NCT02965625
Title: Characterization of Epicardial and Pericardial Adipose Tissue in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other); University of Copenhagen (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Regitse Christensen, MD, Rigshospitalet, Denmark
Other Study IDs: H-16031413
Record Dates: First submitted 2016-10-05; First posted 2016-11-17 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Whole blood Serum Cardiac adipose tissue Cardiac adipose tissue cell culture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- open elective cardiac surgery patients: Including coronary artery bypass graft and valve replacement surgery patients

SUMMARY:
Human epicardial fat is the true visceral fat depot of the heart, and its regional distribution and physiology is of growing scientific and clinical interest. This study aims to characterize the expression profile and function of the epicardial and pericardial adipose tissue compartments of the heart (EAT and PAT). EAT and PAT adipose biopsies will be obtained from patients undergoing coronary artery bypass graft surgery (CABG) or valve replacement surgery.

DETAILED DESCRIPTION:
The epicardial adipose tissue (EAT) stretches from the myocardium to the visceral layer of the pericardium. Adipose located on the outside of the visceral pericardium to the external site of the pericardium is called the pericardial adipose tissue (PAT), and is of a separate origin than EAT. Therefore, this study aims to investigate the global expression profile of the EAT and PAT compartments, in addition to characterizing the function, structure, metabolic and inflammatory profile. Furthermore, this study will determine whether CABG and valve replacement patients display different EAT and PAT characteristics

ELIGIBILITY:
Inclusion Criteria:

* Age <80 years
* Patients undergoing elective heart surgery either for coronary bypass grafting or for other purposes

Exclusion Criteria:

* Inability of the patient to provide informed consent
* Severe kidney failure, GFR<30
* Previous cardio-thoracic surgery
* There are no other specific exclusion criteria, as long as the patient is considered eligible for surgery by the clinicians

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open elective cardiac surgery, specifically coronary artery bypass graft and valve replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Characterization of cardiac adipose tissue | Time of collection during surgery is approximately 3 hours
  Cardiac adipose tissue biopsies will be compared and characterized as brown, beige or white adipose according to gene expression of adipocyte markers

SECONDARY OUTCOMES:
Characterization of cardiac adipose tissue gene expression in coronary artery bypass graft (CABG) and valve replacement surgery patients | Time of collection during surgery is approximately 3 hours
  Gene expression will be measured and compared within cardiac adipose tissue biopsies from patients undergoing CABG or valve replacement surgery.
Characterization of cardiac adipose tissue protein expression in coronary artery bypass graft (CABG) and valve replacement surgery patients | Time of collection during surgery is approximately 3 hours
  Protein expression will be measured and compared within cardiac adipose tissue biopsies from patients undergoing CABG or valve replacement surgery.
Cardiac adipose tissue volume | Prior to surgery
  Cardiac fat volume will be measured by cardiac MRI scan prior to undergoing CABG or valve replacement surgery to assess whether cardiac fat volume correlates with the cardiac adipose profile.
Functional characterization of cardiac adipose biopsy cell culture | Time of collection during surgery is approximately 3 hours
  Primary cell culture will be derived from the cardiac adipose biopsies to perform functional assays in vitro. Gene expression will be measured.
Functional characterization of cardiac adipose biopsy cell culture | Time of collection during surgery is approximately 3 hours
  Primary cell culture will be derived from the cardiac adipose biopsies to perform functional assays in vitro. Protein expression will be measured.
Cardiac muscle biopsies | Time of collection during surgery is approximately 3 hours
  Gene expression in cardiac muscle biopsies and progenitor cells will be compared to that of the adipose biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Regitse H Christensen, MD, Principal Investigator — Rigshospitalet, Denmark; Sarah E Heywood, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Centre for Physical Activity Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No